CLINICAL TRIAL: NCT06536387
Title: Storytelling Through Music: a Novel Approach to Improve Well-being Among Homeless Service Providers
Brief Title: Storytelling Through Music to Improve Well-being Among Homeless Service Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Carolyn Phillips, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00006156
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Burnout, Professional; Anxiety; Depression; Secondary Trauma
Keywords: burnout; music intervention; emotional well-being; work-related stress
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Depression; Compassion Fatigue; Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Storytelling Through Music (Experimental): Storytelling Through Music is a six-week intervention that utilizes storytelling, reflective writing, self-care skills, and song-writing. The intervention will be administered in small groups of 4-6 participants/group and with a hybrid approach. The writing workshops will occur online, and the share circle (stories and songs shared with the group) will occur in person. The group sizes will be kept small to ensure that each participant has adequate time to share their writing during the group sessions.
  Interventions: Behavioral: Storytelling Through Music

INTERVENTIONS:
Behavioral: Storytelling Through Music — Storytelling Through Music is a six-week intervention that combines storytelling, reflective writing, song-writing, and self-care skills to improve emotion regulation through affective and cognitive coping skills.

SUMMARY:
Homelessness is a complex social issue and requires a dedicated workforce of helping professionals, including nurses and social workers. Secondary traumatic stress is common in this workforce and contributes to poor professional quality of life, burnout, and job turnover. These factors undermine the health and well-being of homeless service providers and threaten the stability of this critical workforce. The purpose of this study is to evaluate "Storytelling Through Music," an innovative 6-week, multi-dimensional intervention, to improve well-being among homeless service providers.

DETAILED DESCRIPTION:
Research has found that the burden of secondary traumatic stress among homeless service providers (HSP) is similar to that among other healthcare professionals, including nurses working in urban emergency departments and in inpatient psychiatric hospitals. Left unaddressed, secondary traumatic stress can cause compassion fatigue and emotional exhaustion, furthering a cycle of poor professional quality of life (QoL), burnout, and job turnover. Research has identified that arts-based interventions have promise in helping healthcare professionals cope with work-related emotions, assist in revealing genuine emotions linked to work-related stress, and in improving professional QoL. What remains unclear is if arts-based interventions can yield similar benefits amongst HSPs.

The purpose of this study, therefore, is to evaluate the feasibility of implementing Storytelling Through Music (STM) with HSPs working with the homeless population in Austin, Texas. STM is a six-week intervention that combines storytelling, reflective writing, song-writing, and self-care skills to improve emotion regulation through affective and cognitive coping skills. Our preliminary data suggests STM to be feasible and acceptable, and preliminary evidence demonstrates improved coping, psychosocial well-being, and burnout in nurses. Specifically, this project aims to:

Aim 1: Explore the contextual factors impacting the well-being of frontline HSPs.

Aim 2: Examine the feasibility of implementing Storytelling Through Music with HSPs.

Aim 3: Investigate the preliminary intervention effect on coping (emotion regulation, self-compassion); well-being (anxiety, depressive symptoms, loneliness, post-traumatic growth, insomnia); and work-related factors (secondary traumatic stress, burnout, compassion satisfaction, and intent to leave).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* employed in a homeless services organization in Austin/Travis County for at least 6 months
* licensed as a nurse or social worker
* ability to read and speak English
* access to computer, internet, and zoom.

Exclusion Criteria:

* previous participation in the STM intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Study Feasibility | Immediately post-intervention (6 weeks)
  Feasibility will be evaluated by tracking the percentage of participants screened and enrolled. The study will be deemed feasible with a 60% enrollment rate.
Intervention Feasibility | Immediately post-intervention (6 weeks)
  Feasibility will be evaluated by tracking the average number of sessions the participants complete. This intervention will be deemed feasible if 85% of the intervention is completed.
Intervention Acceptability | Immediately post-intervention (6 weeks)
  An additional primary endpoint is acceptability. Acceptability will be evaluated with semi-structured interview questions to understand the participant's perception of intervention delivery and content, as well as the perceived impact.

SECONDARY OUTCOMES:
Mean Change from Baseline in Anxiety Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short-Form 8a will be used. The minimum score is 8, and the maximum score is 40. Higher scores indicate more anxiety.
Mean Change from Baseline in Depression Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form 8a will be used.The minimum score is 8, and the maximum score is 40. Higher scores indicate higher levels of depressive symptoms.
Mean Change from Baseline in Emotion Regulation Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Trait Emotional Intelligence Questionnaire-Short Form (TEIQue-SF) will be used to assess trait emotional intelligence (EI). The questionnaire consists of 30 items rated on a 7-point scale, provides a global trait EI score, and scores for four subscales (i.e., well-being, self-control, emotionality, and sociability). Higher scores correspond to high levels of trait EI.
Mean Change from Baseline in Self-Compassion Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  Self-Compassion Scale; range is 26-130; higher score is better outcome.
Mean Change from Baseline in Loneliness Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  University of California Los Angeles (UCLA) Loneliness Scale; range is 0-60; lower score is better outcome.
Mean Change from Baseline in Post-traumatic Growth Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Post-traumatic Growth Index (PTGI) consists of 21-items that measures the degree of positive changes in an individual's experience after a challenging life event. The PTGI consists of 5 dimensions: Relating to Others (7-items), New Possibilities (5-items), Personal Strength (4-items), Spiritual Change (2-items), and Appreciation of Life (3-items). Total scores can range from 0 to 105.
Mean Change from Baseline in Insomnia Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short-Form 6a will be used. The minimum score is 6, and the maximum score is 30. Higher scores indicate more sleep disturbance.
Mean Change from Baseline in Professional Quality of Life Scores at 6 weeks and 10 weeks | Immediately post-intervention and 1-month post-intervention
  The Professional Quality of Life (ProQOL) has three subscales: Compassion Satisfaction, Burnout, and Secondary Traumatic Stress. Scores are reported on individual subscales and can range from 10 to 50. Higher levels indicate more of the construct.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Phillips, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No